CLINICAL TRIAL: NCT05981781
Title: Ultrasound Guided Pericapsular Nerve Group Block Versus Ultrasound Guided Caudal Block for Postoperative Pain in Paediatric Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0107623
Record Dates: First submitted 2023-07-10; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain in Paediatric Hip Surgery; PENG Block; Caudal Block
Keywords: PENG block; caudal block; hip surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Double blinded randomized study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the patients , outcome assessors and care providers are not informed with the block type done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided peng block in paediatric hip surgery (Active Comparator): Patients will receive US-guided PENG block with 0.5 ml/kg of bupivacaine 0.25% after induction of general anaesthesia.
  Interventions: Procedure: ultrasound guided peng block in paediatric hip surgery
- ultrasound guided caudal epidural block in paediatric hip surgery (Active Comparator): Patients will receive US-guided caudal block with 0.5 ml/kg of bupivacaine 0.25% after induction of general anaesthesia.
  Interventions: Procedure: ultrasound guided caudal epidural block in paediatric hip surgery

INTERVENTIONS:
Procedure: ultrasound guided peng block in paediatric hip surgery — On the supine position, under strict aseptic technique, a linear, high-frequency transducer (5-13 MHz) of a Sonosite (M-Turbo; Sonosite Inc, Bothell, W, USA) portable US machine will be placed in the transverse plane along the anterior inferior iliac spine (AIIS) to identify the iliopsoas muscle, femoral artery, and femoral nerve. The probe will be then rotated, and aligned with the pubic ramus to visualize the AIIS, iliopubic eminence (IPE), femoral artery, psoas muscle, and the superior pubic ramus.
  Under direct visualization, a needle will be advanced in-plane, lateral to medial between the psoas tendon and pubic ramus until the needle contacts the IPE. The needle will be slightly withdrawn, and following negative aspiration, 0.5 ml/kg of bupivacaine 0.25% will be injected.
  Arms: ultrasound guided peng block in paediatric hip surgery
Procedure: ultrasound guided caudal epidural block in paediatric hip surgery — On lateral decubitus position, under strict aseptic technique, the sacral hiatus will be visualized at the level of the sacral cornua by employing a linear, high-frequency transducer (5-13 MHz) of a Sonosite (M-Turbo; Sonosite Inc, Bothell, W, USA) portable US machine will be placed transversely at the midline to obtain a transverse view of the two cornua, sacrococcygeal ligament, sacral bone, and sacral hiatus. At this level, the ultrasound transducer will be rotated to 90 degree to obtain longitudinal views of the sacrococcygeal ligament and sacral hiatus and subsequently placed between the two cornua. A needle will be advanced toward the upper third of the sacrococcygeal ligament. The needle advancement will be terminated immediately after penetrating the sacrococcygeal ligament. (17) At this level, after confirming absence of blood or cerebrospinal fluid on aspiration, bupivacaine 0.25% (0.5 mL/kg) will be injected over 1 minute while observing an ultrasound longitudinal image.
  Arms: ultrasound guided caudal epidural block in paediatric hip surgery

SUMMARY:
Aim of the study is to evaluate postoperative analgesic effect of ultrasound guided PENG block in comparison to ultrasound guided caudal epidural anaesthesia for hip surgeries in paediatrics

DETAILED DESCRIPTION:
Hip surgeries in paediatric patients such as open hip surgery for correction of developmental dysplasia of the hip (DDH) lead to extensive injuries and severe pain. Multimodal analgesia is required to provide intraoperative and postoperative analgesia and to prevent the undesirable side effects of opioids including sedation, nausea, vomiting and constipation.

Perioperative pain control is of paramount importance during paediatric hip surgery. Inadequate analgesia can contribute to patient and parental dissatisfaction, prolonged recovery, and increased length of hospital stay. As such, regional anaesthesia is advantageous in providing sufficient analgesia while reducing the adverse effects of opioids. The use of regional anaesthesia in the paediatric population has increased over the last decade as it offers several potential advantages in the provision of postoperative analgesia including a reduction in parenteral opioids, decreased exposure to general anaesthetic agents, and shortened hospital stay. Such techniques may be particularly valuable following painful orthopedic procedures including hip and femur surgery.

Neuraxial techniques (caudal and intrathecal), lumbar plexus blockade, and combined femoral nerve and fascia iliaca blockade have been shown in a myriad of paediatric studies to exhibit opioid-sparing effects and lower postoperative pain scores in patients who are suffering from hip pain.

Caudal block is a common technique used for perioperative pain relief in paediatric lower limb surgeries but despite the success of neuraxial blocks in decreasing postoperative pain scores in paediatric patients undergoing hip surgery, positioning requirements, bilateral sensory and motor blockade, and urinary retention limit their use.

Among peripheral nerve block techniques used for relieving pain associated with hip fracture, ultrasound-guided femoral nerve (FN) block, fascia iliaca compartment (FIC) block and 3-in-1 FN block are widely used. However, these techniques have often failed to provide adequate block of the obturator nerve (ON) and the accessory obturator nerve (AON).

The pericapsular nerve group (PENG) block is an ultrasound guided approach, first described by Girón-Arango et al.(11) in 2018 for the anaesthetizing the articular branches of the femoral, obturator and accessory obturator nerves that provide sensory innervation to the anterior hip capsule. It is a plane block involving one injection, performed under ultrasound guidance, of a high volume of local anaesthetic into the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. It was suggested that the articular branches of ON were blocked successfully due to the proximity of the target area to the subpectineal plane.

PENG block has been initially used as an alternative regional anaesthetic technique for the management of acute pain after hip fracture , but its applications are expanding, suggesting a potential role for analgesia after elective hip surgery. Previous studies concluded that this technique could provide an effective blockade of the articular branches of FN, ON and AON, with a potential motor-sparing effect.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients belonging to American society of anesthesiologists (ASA)class1 or 2, aged 2-8 years scheduled for hip surgery

Exclusion Criteria:

* parent refusal skin infection at site of injection bleeding disorder or receiving anticoagulants history of allergy or contraindicaion to local anaesthetics neurological disease as cerebral palsy

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | 24 hours
  compare between both groups as regard postoperative opioid consumption

SECONDARY OUTCOMES:
postoperative analgesia | 24 hours
  postoperative analgesia by using FLACC scale
duration of postoperative analgesia | 24 hours
heamodynamics | 24 hours
  changes in heart rate
incidence of complications | 24 hours
  hypotension, bradycardia, nausea, vomiting, urinary retention, and pruritis
parent satisfaction | 24 hours
  Using a 5 point score (0= very dissatisfied, 1= dissatisfied, 2= neither satisfied nor dissatisfied, 3= satisfied, 4= very satisfied)

OTHER OUTCOMES:
heamodynamics | 24 hours
  Changes in arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Rabab Saber, professor, Study Director — Alexandria University; Aly Mahmoud, lecturer, Study Director — Alexandria University; Ahmed Mansour, professor, Study Director — Alexandria University; yomna Said, MBBCH, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data results and statistical analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: before the start till publishing the study
Access Criteria: not public only researchers who can access study information